CLINICAL TRIAL: NCT07367854
Title: Impact of Food Combinations on the Stimulation of Post-exercise Muscle Protein Synthesis in Healthy Adults
Brief Title: Diet Synergy in Muscle Protein Synthesis
Acronym: POTATO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Nicholas Burd, Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-1113; UI Award #123640 (Other Grant/Funding Number: Nutrition in Demand)
Record Dates: First submitted 2025-12-04; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Muscle Protein Synthetic Response to Protein; Muscle Protein Synthesis; Muscle Health; Protein Metabolism; Recreational Activities; Isotope Labeling
Keywords: protein; leucine kinetics; food matrix; protein synthesis; potato; stable isotope tracers; constant infusions; food combinations
MeSH Terms: interventions — Resistance Training; Red Meat; Bread

STUDY DESIGN:
Intervention Model Description: Randomized semi-crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Potato and Beef (PB) (Experimental): Participants will ingest 1 medium russet potato with skins and 2 ounce-equivalent lean ground beef combination (274 kcals, 19.3 g protein, 37 g carbohydrate, 5 g fat, 4 g fiber) after resistance exercise.
  Interventions: Behavioral: Resistance Exercise; Dietary Supplement: Potato and Beef
- Bread and Beef (BB) (Experimental): Participants will ingest 2 slices white bread and 2 ounce-equivalent lean ground beef combination (262 kcals, 19.8 g protein, 28 g carbohydrate, 6.8 g fat, 1.8 g fiber) after resistance exercise.
  Interventions: Behavioral: Resistance Exercise; Dietary Supplement: Bread and Beef
- Beef (B) (Experimental): Participants will ingest 2 ounce-equivalent lean ground beef (110 kcals, 14.8 g protein, 5 g fat) after resistance exercise.
  Interventions: Behavioral: Resistance Exercise; Dietary Supplement: Beef

INTERVENTIONS:
Behavioral: Resistance Exercise — Participants will perform leg press and leg extension immediately prior to ingestion of either potato-beef combination, bread-beef combination, or beef alone.
Dietary Supplement: Potato and Beef — Participants will ingest baked russet potato and cooked ground beef immediately after resistance exercise.
  Arms: Potato and Beef (PB)
Dietary Supplement: Bread and Beef — Participants will ingest white bread and cooked ground beef immediately after resistance exercise.
  Arms: Bread and Beef (BB)
Dietary Supplement: Beef — Participants will ingest cooked ground beef immediately after resistance exercise.
  Arms: Beef (B)

SUMMARY:
In the present semi-crossover randomized design, 15 recreationally active young adults (19-40 y) will receive stable isotope tracer infusions and perform a single bout of resistance exercise. Immediately after exercise, participants will ingest either 1 medium russet potato with skins and 2 ounce-equivalent lean ground beef combination (274 kcals, 19.3 g protein, 5 g fat, 37 g carbohydrates, and 4 g fiber), 2 slices of white bread and beef combination (262 kcals, 19.8 g protein, 6.8 g fat, 28 g carbohydrates, and 1.8 g fiber) or 2 ounce-equivalent beef (93% lean meat/7% fat; 110 kcals, 14.8 g protein, and 5 g fat). Repeated blood and muscle biopsies will be collected to determine whole body leucine kinetics, amino acid concentrations, anabolic signaling and myofibrillar protein synthesis rates during the trials.

DETAILED DESCRIPTION:
1. Preliminary Testing

   1.1 Preparations: Participants will arrive for the preliminary testing session after an overnight fast (~10 h no caloric foods/beverages consumed) and having refrained from exercise for the 72 h prior. Prior to any in-person procedures, participants will be briefed on the procedures and risks associated with participation via reviewing the informed consent document. Participants will be encouraged to ask questions and have their questions answered prior to being asked if they'd like to continue. Confirmation will be documented via signature on an informed consent process form.

   1.2 Anthropometrics: Upon provision of consent, participants' height and weight will be measured to confirm body mass index (BMI) is within eligibility limits (18.5 - 30 kg/m^2). Since participants have already been assessed for all other inclusion and exclusion criteria, an eligible BMI will result in study inclusion and continuation of the preliminary testing session. Following confirmation of study eligibility, blood pressure will be measured by a trained member of the research team. Subsequently, body composition will be determined via dual energy x-ray absorptiometry (DEXA) in accordance with manufacturer recommendations. Briefly, participants will be asked to remove all metal objects from their person prior to being positioned by a trained technician for accurate measurement of lean body mass and fat mass. The scan lasts approximately 6-10 minutes during which the participant will be instructed to remain motionless.

   1.3 Habitual Diet Record: Current diet habits will be assessed through an online automated self-administered (ASA24) diet record system. Participants will receive their individual username and password during this session and will be asked to record for 3 consecutive days (2 weekdays and 1 weekend day) prior to each trial. Since it is online, participants can complete it off-site at their leisure.

   1.4 Resting Metabolic Rate: Resting metabolic rate (RMR) will be assessed via indirect calorimetry. This is a non-exertional test whereby RMR is measured using an automated gas analysis system. This device measures oxygen consumption and carbon dioxide production as the difference between inspired and expired gas concentrations. Prior to the beginning of the test, participants will lie supine on a table and a clear, hard plastic hood and soft, clear plastic drape will be placed over the participants neck, head, and shoulders to capture expired gases. Participants will then lie motionless without falling asleep while respiratory gas concentrations are captured. Testing will conclude when RMR is stable for at least 20 min (typically ~30 min from the onset).

   1.5 Ten-Repetition Maximum (10RM) Testing: Following resting metabolic rate testing, participants will have their 10RM tested for the leg extension and leg press. To begin, participants will cycle at a self-selected pace on a standard cycle ergometer for ~5 minutes. Participants will then complete a set of 8-10 repetitions at ~50% of their predicted 10RM followed by 1-2 minutes of rest. The load will then be set at ~90% of their predicted 10RM. Load will be increased by 2.5-5.0% following each successful attempt until failure (typically within 5 attempts). Two minutes of rest will be allotted between maximal attempts and 5 minutes between exercises. Leg extension will be tested first followed by leg press. Before leaving the laboratory, participants will be allowed to ask any questions they have before concluding the session.

   1.6 Accelerometers: Prior to leaving the laboratory, participants will be given an accelerometer (Actigraph) to assess levels of daily physical activity (i.e step count). Research personnel will demonstrate proper use and instruct participants to wear the device throughout the entire duration of the study. Following the demonstration, participants will be reminded to refrain from any extraneous exercise and wear the device for two days leading into the trials.

   1.7 Planning: Prior to leaving the laboratory, participants and the research team will identify a date for the first infusion trial (at least 7 days following preliminary testing). Moreover, the research team will provide participants with a standardized meal to consume the night before the first infusion and instructions to refrain from strenuous exercise and alcohol consumption for 72 and 24 hours leading into the first trial. Participants will also be offered a snack prior to leaving the laboratory.
2. Infusion Trials

2.1 Preparations: At least 7 days following preliminary testing or the previous infusion, participants will be asked to return to the laboratory for an infusion trial. On the morning of each infusion, participants will arrive to the laboratory in the morning following an overnight (~10 h no caloric foods/beverages consumed) fast and having refrained from strenuous exercise and alcohol consumption for 72 and 24 hours, respectively. For 3 days preceding each trial, participants will be asked to record their dietary intakes via and online automated self-administered (24 hour) dietary record system (ASA24).

2.2 Stable Isotope Infusion: Upon arrival to the laboratory, participants will lay supine on a clinic-style bed before having an intravenous catheter placed into a dorsal hand or arm vein. No more than four attempts will be made to set the catheter. Following baseline blood sampling, a priming dose of L-[1-13C] leucine and L-[ring 2H5] phenylalanine will be administered prior to initiation of a constant infusion using a calibrated infusion pump. The stable isotope amino acid tracers applied in this experiment are not radioactive and are completely safe. These stable isotopes will enrich the amino acid pool in the body allowing us to identify the rate of incorporation of amino acids into the tissues. The preparation of the tracers for intravenous administration will occur in a sterile environment under a laminar flow hood dedicated to the preparation of tracers and in accordance with Good Manufacturing Practices guidelines.

2.3 Blood Collection: After investigators start the infusion, a second catheter will be placed in a hand or arm vein on the other side so investigators can collect blood throughout the trial. Throughout the trial, blood will be collected periodically from the catheter. Before the collection of some samples, a heated blanket (60°C) will be placed on the catheter site (arm or hand) to "arterialize" (mimic the blood within arteries) the blood samples. A total of 17 blood samples (~174 mL) will be collected during the first trial, while in the second trial, 15 blood samples (~149 mL) will be collected. The regular collection of blood allows the determination of the isotopic enrichment, amino acid concentrations and free fatty acid concentrations in blood. Between draws, the catheter will be kept patent using a 0.9% saline drip at a low rate.

2.4 VCO2: Carbon dioxide production (VCO2) will be determined from expired air sampled by open circuit mouthpiece attached to a hose. Immediately after VCO2 analysis is performed (10 minutes), participants will be asked to exhale into a separate mouthpiece attached to a plastic bag. This breath sample is stored in a sterile vacutainer for future analysis of stable isotope tracer enrichment in the breath.

2.5 Muscle Collection: A total of five muscle biopsies will be collected (three as a part of 1st infusion and two during 2nd infusion). The biopsy procedure involves removal of a small piece of muscle tissue using a sterile hollow needle (Bergström needle) and will be performed by Dr. Nicholas Burd under the auspices of Dr. Jared Willard, MD. Participants will rest on a bed and the area for the biopsy will be shaved, if required. Subsequently, the area will be sterilized using 4% chlorhexidine gluconate before 5 mL of local anesthetic (2% Xylocaine with 1:100,000 epinephrine) is injected subcutaneously with special care to avoid infiltrating the muscle. Once the anesthetic is active (~10 min), Dr. Burd will make a small incision (~4-5 mm) in the skin in order to create an opening through which to put the biopsy needle for tissue collection. Dr. Burd will quickly cut of a small piece of muscle (~50- 100 mg; about the size of a standard pencil eraser) and remove the needle from the subject's leg. During the sample collection (~30 sec), the subjects may feel a sensation of deep pressure in their leg. A sterile disposable drape will be placed under the participant's thigh and sterile gloves will be used for all biopsy procedures.

After the biopsy is completed, a trained research team member will apply pressure with sterile gauze until the bleeding stops (at least 10 min). Subsequently, the incision site will be closed using butterfly stitches (Steri-strips) following by application of a bandage. An elastic pressure wrap will be applied on top of the bandage in order to minimize the chance of bruising. Participants will then be instructed to leave the butterfly stitches and the pressure wrap on the wound for 96 and 24 hrs, respectively. The participant will be provided with a "biopsy care kit" (described in section 10.1/Biopsy care kit) in order to properly care for the incision after leaving the laboratory. A member of the research team will contact the participants in the day following the trial to check on the healing process.

Resistance Exercise and Meal Ingestion: Immediately following closure of the second biopsy, participants will begin warming up for an acute bout of resistance exercise. To begin, participants will cycle at a self-selected pace on a standard cycle ergometer for 5 minutes. Subsequently, participants will begin resistance exercise. Participants will complete a warmup set at ~60% of their ten-repetition maximum (10RM) measured at preliminary testing followed by 4 sets of 10-12 repetitions at ~90% 10RM with 1-3 minutes rest between sets for both leg extension and leg press. Participants will match the load, sets, and repetitions from the first trial during their second trial.

Immediately following the completion exercise, participants will return to the infusion room to consume meals. During first trial, participants will be randomized and counterbalanced to ingest either 1 medium russet potato with skins and 2 ounce-equivalent lean ground beef combination (274 kcals, 19.3 g protein, 5 g fat, 37 g carbohydrates, and 4 g fiber), 2 slices white bread and beef combination (262 kcals, 19.8 g protein, 6.8 g fat, 28 g carbohydrates, and 1.8 g fiber), or 2 ounce-equivalent beef (93% lean meat/7% fat; 110 kcals, 14.8 g protein, and 5 g fat) during the primed constant infusions for the measurement of protein metabolism. During second trial, participants will be randomly assigned to consume one of the remaining conditions.

Commercially available russet potato with skins will be cut into 1-inch cubes and baked alongside ground beef patty at 200°C for ~30 minutes, or until the internal temperature of the beef reaches 75°C right before consumption on the trial day. The meal will be cooked to an internal temperature of at least 165°F in accordance with the USDA's minimum internal temperature to prevent foodborne illness.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-40 yrs
* Pre-menopausal
* Recreationally-active
* Weight stable for prior 6 months

Exclusion Criteria:

* Age outside of range (20 - 35 yrs)
* Pregnancy
* Irregular menstrual cycles (i.e., ~21 day or ~35 day cycle)
* Participation in previous research using L-[1-13C] leucine and L-[ring-2H5] phenylalanine
* Participation in other ongoing research that interferes with this study (e.g., conflicting diet, activity interventions, etc.)

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-03-03 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Myofibrillar protein fractional synthesis rate | Baseline muscle biopsy (-150 minutes), Postabsorptive muscle biopsy (-30 minutes), and Postprandial muscle biopsy (300 minutes)
  Myofibrillar protein synthesis rates will be assessed during the postabsorptive and postprandial periods of experimental primed-constant stable isotope infusions.
Whole body leucine kinetics | Breath sample collection time points: -210, -150, -90, -60, -30, 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240, and 300 minutes.
  Whole body leucine kinetics will be determined via breath sample collection during the postabsorptive and postprandial periods of experimental primed-constant stable isotope infusions and analyzed via LC/MS/MS.

SECONDARY OUTCOMES:
Activation of anabolic signaling targets | Baseline muscle biopsy (-150 minutes), Postabsorptive muscle biopsy (-30 minutes), and Postprandial muscle biopsy (300 minutes)
  Phosphorylation of mTOR-dependent anabolic signaling targets (i.e., 4E-BP1, S6K1, and rps) will be assessed via Western Blotting (phosphorylated-to-total ratio).

CONTACTS AND LOCATIONS:
Locations (1):
- Louise Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Because it is not planned to published in any ICMJE journal.